CLINICAL TRIAL: NCT00324207
Title: Prediction of Type 1 Diabetes: Molecular Quantification of Insulin mRNA in the While Cell Fraction of Whole Blood
Brief Title: Molecular Quantification of Insulin mRNA
Status: Completed | Type: Observational
Sponsor: Children's Mercy Hospital Kansas City (Other)
Responsible Party: Wayne Moore, MD, PhD, The Children's Mercy Hospital
Other Study IDs: 00006028; 00006028
Record Dates: First submitted 2006-05-08; First posted 2006-05-10 (Estimated); Last update posted 2010-03-05 (Estimated); Status verified 2010-03

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: Type 1 diabetes mellitus; Insulin mRNA
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The objectives of this study are to:

1. quantitate the level of insulin mRNA in the while cell fraction of whole blood in selected groups of subjects,
2. determine the gene expression of markers of white cell activation in the white cell fraction of whole blood in selected subjects,
3. determine the identity of the white cell responsible for expression of insulin mRNA and
4. determine protein expression of mRNA of insulin/proinsulin and selected genes of white cell activation.

DETAILED DESCRIPTION:
Indicators of active immune or chemically mediated beta cell destruction would be helpful for predicting the development and severity of autoimmune diabetes and monitoring the success of islet transplants. Currently there are no reliable indicators readily available.

Insulin mRNA in the white cell fraction of blood has been detected or elevated under several circumstances including:

1. normal animals
2. after islet cell transplantation
3. hyperglycemic induced expression and
4. during induction of diabetes with streptozotocin

The investigators propose that quantitative measurement of insulin mRNA may be an accurate, innovative and minimally invasive indicator of beta cell destruction.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects ages 1 to 17 years of age
2. Subjects with evidence of beta cell dysfunction or evidence of beta cell autoimmunity
3. Subjects with new onset type 1 diabetes
4. Non-diabetic and autoantibody negative siblings of subjects with new onset type 1 diabetes
5. Unrelated nondiabetic controls with no family history of type 1 diabetes
6. Of sufficient size to donate 10ml of blood

Exclusion Criteria:

None if subjects meet above inclusion criteria

Ages: 1 Year to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Hospital and clinic patients and their siblings.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2006-02; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wayne Moore, MD, PhD, Principal Investigator — Children's Mercy Hospital Kansas City
Locations (1):
- Children's Mercy Hospital, Kansas City, Missouri, United States